CLINICAL TRIAL: NCT00635804
Title: A 2-Part, Randomized, Double-Blind, Placebo-Controlled, Multiple-Rising Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MK-3281 in Healthy Male Subjects and Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-3281 in Hepatitis C Infected Male Patients
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MK-3281 in Healthy and Hepatitis C Infected Male Participants (MK-3281-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3281-002; 2008_507 (Other: Merck Registration Number); 2007-006245-40 (EudraCT Number)
Record Dates: First submitted 2008-02-28; First posted 2008-03-14 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — 14-cyclohexyl-7-((2-(dimethylamino)ethyl)(methyl)amino)-7,8-dihydro-6H-indolo(1,2-e)(1,5)benzoxazocine-11-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Pt 1: MK-3281 100 mg BID (Panel A) (Experimental): Healthy male participants in this Part I serial panel receive 100 mg MK-3281 orally twice daily (BID) for 10 consecutive days for a total daily dose administered of 200 mg. The evening (PM) dose of MK-3281 was not administered on Day 10.
  Interventions: Drug: MK-3281
- Pt 1: MK-3281 200 mg BID (Panel B) (Experimental): Healthy male participants in this Part I serial panel receive 200 mg MK-3281 orally BID for 10 consecutive days for a total daily dose administered of 400 mg. The PM dose of MK-3281 was not administered on Day 10.
  Interventions: Drug: MK-3281
- Pt 1: MK-3281 400 mg BID (Panel C) (Experimental): Healthy male participants in this Part I serial panel receive 400 mg MK-3281 orally BID for 10 consecutive days for a total daily dose administered of 800 mg. The PM dose of MK-3281 was not administered on Day 10.
  Interventions: Drug: MK-3281
- Pt 1: MK-3281 800 mg BID (Panel D) (Experimental): Healthy male participants in this Part I serial panel receive 800 mg MK-3281 orally BID for 10 consecutive days for a total daily dose administered of 1600 mg. The PM dose of MK-3281 was not administered on Day 10.
  Interventions: Drug: MK-3281
- Pt 2: MK-3281 800 mg BID (Panel E) (Experimental): Genotype (GT)1 HCV-infected male participants in this Part II serial panel receive 800 mg MK-3281 orally BID for 7 consecutive days for a total daily dose administered of 1600 mg. The PM dose of MK-3281 was not administered on Day 7.
  Interventions: Drug: MK-3281
- Pt 2: MK-3281 800 mg BID (Panel F) (Experimental): GT1a/GT1-nontypeable/GT3/GT1b HCV-infected male participants in this Part II serial panel receive 800 mg MK-3281 orally BID for 7 consecutive days for a total daily dose administered of 1600 mg. The PM dose of MK-3281 was not administered on Day 7.
  Interventions: Drug: MK-3281
- Pt 2: MK-3281 1200 mg BID (Panel G) (Experimental): GT1a (and/or GT1 nontypeable) and GT1b HCV-infected male participants in this Part II serial panel receive 1200 mg MK-3281 orally BID for 7 consecutive days for a total daily dose administered of 2400 mg. The PM dose of MK-3281 was not administered on Day 7.
  Interventions: Drug: MK-3281
- Placebo (Placebo Comparator): Participants receive dose-matched placebo to MK-3281 orally BID for 7 or 10 consecutive days depending on randomization. The PM dose of matched placebo was not administered on Day 7 or 10 (depending upon allocation).
  Interventions: Drug: Placebo to MK-3281

INTERVENTIONS:
Drug: MK-3281 — MK-3281 capsule administered orally BID for 7 or 10 consecutive days depending on randomized dose. The PM dose of MK-3281 was not administered on Day 7 (for HCV-infected males) or Day 10 (for healthy males)
  Arms: Pt 1: MK-3281 100 mg BID (Panel A); Pt 1: MK-3281 200 mg BID (Panel B); Pt 1: MK-3281 400 mg BID (Panel C); Pt 1: MK-3281 800 mg BID (Panel D); Pt 2: MK-3281 1200 mg BID (Panel G); Pt 2: MK-3281 800 mg BID (Panel E); Pt 2: MK-3281 800 mg BID (Panel F)
Drug: Placebo to MK-3281 — Dose-matched placebo to MK-3281 capsule administered orally BID for 7 or 10 consecutive days depending on randomized dose of MK-3281 in serial panel. The PM dose of matched placebo was not administered on Day 7 or 10 (depending upon allocation).
  Arms: Placebo

SUMMARY:
This study will examine the safety, tolerability and plasma pharmacokinetics of multiple doses of MK-3281 in healthy male participants in Part I, and in Hepatitis C Virus (HCV)-infected male participants in Part II. The clinical efficacy of MK-3281, as measured by viral load reduction, will also be assessed in Part II. The primary hypothesis is that twice daily administration of MK-3281 for 10 days in healthy adult male participants and for 7 days in HCV-infected male participants is sufficiently safe and well tolerated, based on assessment of clinical and laboratory adverse experiences, to permit continued clinical investigation.

The results of this study will guide dose selection for future studies in both healthy participants and HCV-infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged to be in good/stable health based on medical history, physical examination, vital signs, and laboratory safety tests performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug
* Participant has no clinically significant abnormality on electrocardiogram (ECG) performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug
* Participants with female partner(s) of childbearing potential must agree to use a medically acceptable method of contraception during the study and for 90 days after the last dose of study drug
* Participant has a clinical diagnosis of chronic HCV infection (for Part II only).

Exclusion Criteria:

* Participant has a history of stroke, chronic seizures, or major neurological disorder
* Participant has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Participant has a history of neoplastic disease (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment
* Participant has positive Hepatitis B surface antigen (or other evidence of active Hepatitis B infection) at the prescreening (study) visit
* For Healthy Panel (Part I), participant has evidence of chronic Hepatitis C virus infection at the prescreening (study) visit
* Participant has a history of documented Human Immunodeficiency Virus (HIV) infection

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02-19 (Actual); Primary Completion 2009-12-22 (Actual); Study Completion 2009-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3281-002&kw=3281-002&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Panel H, planned for GT1a/GT1b HCV-infected male participants to receive 400 mg MK-3281 orally BID for 7 consecutive days, did not enroll any participants. As pre-specified by the protocol, it was possible that some panels would not be enrolled if study objectives were met with prior doses.
Pre-assignment Details: 60 participants were enrolled in this study and received MK-3281 or placebo in Panels A through G.
Groups:
- Pt 2: MK-3281 800 mg BID (Panel E): Genotype (GT)1 Hepatitis C Virus (HCV)-infected male participants in this Part II serial panel received 800 mg MK-3281 orally BID for 7 consecutive days for a total daily dose administered of 1600 mg. The PM dose of MK-3281 was not administered on Day 7.
- Placebo: Participants receive dose-matched placebo to MK-03281 orally BID for 7 or 10 consecutive days depending on randomization. The PM dose of matched placebo was not administered on Day 7 or 10 (depending upon allocation).
Period: Overall Study
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Started | 7 | 6 | 6 | 6 | 6 | 12 | 3 | 14
Completed | 6 | 6 | 6 | 6 | 6 | 11 | 3 | 14
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 12 | 3 | 14 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (8.7) | 36.3 (13.5) | 37.0 (13.0) | 34.0 (14.9) | 39.2 (7.3) | 47.5 (8.8) | 45.0 (5.2) | 39.4 (10.0) | 39.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 6 | 6 | 6 | 6 | 12 | 3 | 14 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, was also an AE.
Time Frame: Up to 14 days after the last dose of study drug (up to 24 days maximum)
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 12 | 3 | 14
participants | 5 | 3 | 4 | 5 | 3 | 12 | 2 | 12

2. Primary Outcome: Number of Participants Who Discontinued Study Medication Due to AEs
Description: as for outcome 1
Time Frame: Up to 14 days after the last dose of study drug (up to 24 days maximum)
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 12 | 3 | 14
participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Time 12 Hours (AUC[0-12]) of MK-3281
Description: Blood samples were obtained from participants and MK-3281 AUC(0-12) was calculated at Days 1 and 7 (for HCV+ participants) or Day 10 (for healthy participants) using the MK-3281 assay.
Time Frame: Predose daily on Days 2-9 (for healthy participants) and Days 2-6 (for HCV+ participants), and predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose on Day 1, Day 7 (HCV+ participants), and Day 10 (healthy participants)
Population: All Treated Participants with available PK data. Participants in the Placebo group did not receive MK-3281 and therefore did not have PK data reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
μM·hr
  Day 1 | 4.92 (39.9) | 12.39 (36.2) | 13.21 (45.0) | 18.12 (70.9) | 12.78 (22.4) | 11.36 (47.7) | 12.01 (27.5) |
  Day 7 | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | 61.08 (20.1) | 51.68 (29.8) | 88.21 (37.0) |
  Day 10 | 11.51 (31.7) | 29.71 (32.1) | 37.21 (22.6) | 67.11 (28.1) | NA (NA) — This group did not receive MK-3281 on this day. | NA (NA) — This group did not receive MK-3281 on this day. | NA (NA) — This group did not receive MK-3281 on this day. |

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-3281
Description: Blood samples were obtained from participants and MK-3281 Cmax was calculated at Days 1 and 7 (for HCV+ participants) or Day 10 (for healthy participants) using the MK-3281 assay.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
μM
  Day 1 | 0.74 (32.6) | 1.75 (39.1) | 1.80 (48.3) | 2.73 (75.9) | 1.61 (24.9) | 1.60 (43.7) | 1.69 (28.4) |
  Day 7 | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | 6.78 (23.9) | 5.60 (33.3) | 10.73 (40.5) |
  Day 10 | 1.28 (28.3) | 3.45 (36.2) | 4.97 (44.1) | 7.83 (48.8) | NA (NA) — This group did not receive MK-3281 on this day. | NA (NA) — This group did not receive MK-3281 on this day. | NA (NA) — This group did not receive MK-3281 on this day. |

5. Secondary Outcome: 12-Hour Concentration of MK-3281 in Plasma (C12hr)
Description: Blood samples were obtained from participants and MK-3281 plasma C12hr was calculated at Days 1 and 7 (for HCV+ participants) or Day 10 (for healthy participants) using the MK-3281 assay.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
μM
  Day 1 | 0.26 (42.3) | 0.61 (35.2) | 0.70 (40.5) | 0.95 (73.1) | 0.76 (29.7) | 0.64 (66.1) | 0.64 (26.6) |
  Day 7 | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | 3.62 (25.7) | 3.09 (26.9) | 4.90 (32.1) |
  Day 10 | 0.64 (40.3) | 1.66 (32.1) | 1.86 (26.3) | 2.87 (24.2) | NA (NA) — This group did not receive MK-3281 on this day. | NA (NA) — This group did not receive MK-3281 on this day. | NA (NA) — This group did not receive MK-3281 on this day. |

6. Secondary Outcome: Time To Reach Cmax (Tmax) of MK-3281
Description: Blood samples were obtained from participants and MK-3281 Tmax was calculated at Days 1 and 7 (for HCV+ participants) or Day 10 (for healthy participants) using the MK-3281 assay.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
hour
  Day 1 | 3.0 (42.3) [1.5 to 6.0] | 2.0 (35.2) [1.5 to 3.0] | 5.0 (40.5) [3.0 to 6.0] | 3.0 (73.1) [1.5 to 4.0] | 2.5 (29.7) [1.4 to 4.0] | 3.0 (66.1) [1.5 to 6.0] | 3.0 (26.6) [3.0 to 3.1] |
  Day 7 | NA (NA) [NA to NA] — This group was not assessed for PK on this day. | NA (NA) [NA to NA] — This group was not assessed for PK on this day. | NA (NA) [NA to NA] — This group was not assessed for PK on this day. | NA (NA) [NA to NA] — This group was not assessed for PK on this day. | 2.3 (25.7) [0.0 to 2.8] | 2.0 (26.9) [1.0 to 3.0] | 1.0 (32.1) [0.0 to 1.5] |
  Day 10 | 3.5 (40.3) [2.0 to 4.0] | 3.0 (32.1) [2.0 to 4.0] | 3.5 (26.3) [1.5 to 6.0] | 3.0 (24.2) [1.5 to 4.0] | NA (NA) [NA to NA] — This group did not receive MK-3281 on this day. | NA (NA) [NA to NA] — This group did not receive MK-3281 on this day. | NA (NA) [NA to NA] — This group did not receive MK-3281 on this day. |

7. Secondary Outcome: Apparent Half-Life (t ½) of MK-3281
Description: Blood samples were obtained from participants and MK-3281 apparent t ½ was calculated at Day 7 (for HCV+ participants) or Day 10 (for healthy participants) using the MK-3281 assay. Harmonic mean t ½ and pseudo standard deviation were reported.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours post-dose on Day 7 (HCV+ participants) or Day 10 (healthy participants)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
hour
  Day 7 | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | NA (NA) — This group was not assessed for PK on this day. | 18.3 (4.0) | 19.7 (3.3) | 19.5 (2.0) |
  Day 10 | 17.2 (2.3) | 17.5 (2.9) | 17.4 (2.5) | 16.9 (1.3) | NA (NA) — This group did not receive MK-3281 on Day 10, thus this day was not used to calculate t 1/2. | NA (NA) — This group did not receive MK-3281 on Day 10, thus this day was not used to calculate t 1/2. | NA (NA) — This group did not receive MK-3281 on Day 10, thus this day was not used to calculate t 1/2. |

8. Secondary Outcome: AUC (0-12hr) Accumulation Ratio of MK-3281
Description: Blood samples were obtained from participants and the MK-3281 AUC(0-12hr) accumulation ratio was calculated for HCV+ participants and healthy participants. AUC(0-12hr) accumulation ratio calculated for healthy participants as Day 10 AUC (0-12hr) / Day 1 AUC (0-12hr). AUC(0-12hr) accumulation ratio calculated for HCV+ participants as Day 7 AUC (0-12hr) / Day 1 AUC (0-12hr).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
ratio | 2.3 (NA) [1.6 to 3.4] | 2.4 (NA) [1.6 to 3.5] | 2.8 (NA) [1.9 to 4.1] | 3.7 (NA) [2.5 to 5.6] | 4.8 (4.0) [3.6 to 6.4] | 4.5 (3.3) [3.7 to 5.6] | 7.3 (2.0) [4.9 to 11.1] |

9. Secondary Outcome: Cmax Accumulation Ratio of MK-3281
Description: Blood samples were obtained from participants and the MK-3281 Cmax accumulation ratio was calculated for HCV+ participants and healthy participants. Cmax accumulation ratio calculated for healthy participants as Day 10 Cmax / Day 1 Cmax. Cmax accumulation ratio calculated for HCV+ participants as Day 7 Cmax / Day 1 Cmax.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
ratio | 1.7 (NA) [1.2 to 2.6] | 2.0 (NA) [1.3 to 3.0] | 2.8 (NA) [1.8 to 4.2] | 2.9 (NA) [1.9 to 4.4] | 4.2 (4.0) [3.0 to 5.9] | 3.5 (3.3) [2.7 to 4.4] | 6.4 (2.0) [4.0 to 10.1] |

10. Secondary Outcome: C12hr Accumulation Ratio of MK-3281
Description: Blood samples were obtained from participants and the MK-3281 C12hr accumulation ratio was calculated for HCV+ participants and healthy participants. C12hr accumulation ratio calculated for healthy participants as Day 10 C12hr / Day 1 C12hr. C12hr accumulation ratio calculated for HCV+ participants as Day 7 C12hr / Day 1 C12hr.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 3 | 0
ratio | 2.5 (NA) [1.6 to 4.1] | 2.7 (NA) [1.7 to 4.4] | 2.6 (NA) [1.6 to 4.3] | 3.0 (NA) [1.9 to 4.9] | 4.7 (4.0) [3.6 to 6.2] | 4.8 (3.3) [4.0 to 5.8] | 7.7 (2.0) [5.3 to 11.2] |

11. Secondary Outcome: Maximum HCV Viral Load Change From Baseline Over Study Following MK-3281 Dosing For 7 Days
Description: For evaluation of MK-3281 antiviral activity, the maximum reduction in HCV ribonucleic acid (RNA) levels over the course of the study was assessed by MK-3281 dose group in HCV+ participants and the mean maximum viral load reduction was summarized. HCV RNA levels were measured at predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 hours postdose on Day 1 and Day 7; pre-morning (AM) and pre-evening (PM) dose Day 2; and pre AM dose Days 3-6. For each participant, baseline measurement was defined as the measurement obtained pre-dose on the first day of dosing, and change from baseline (difference) was calculated at each time point. The response for that participant was defined as: - (postbaseline time point - baseline) at the time point with the lowest HCV RNA level.
Time Frame: Baseline (pre-dose Day 1), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
Population: Treated HCV+ participants in Part II with available HCV RNA data. 800 mg dose group contained members of Panels E and F. No healthy participants from Part 1 (Panels A, B, C, or D) were assessed for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: log(IU/ml)
Groups:
- Pt 2: MK-3281 800 mg BID (Panels E+F): GT1/GT1a/GT1-nontypeable/GT3/GT1b HCV-infected male participants receive 800 mg MK-3281 orally BID for 7 consecutive days for a total daily dose administered of 1600 mg. The PM dose of MK-3281 was not administered on Day 7.
- Placebo: HCV-infected participants in Part II who received dose-matched placebo to MK-03281 orally BID for 7 consecutive days.
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panels E+F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 17 | 3 | 6
log(IU/ml) |  |  |  |  | 1.95 [1.36 to 2.54] | 1.34 [-0.34 to 3.01] | 0.37 [0.20 to 0.54]

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug (up to 24 days maximum)
Description: AEs were reported for All Treated Participants.
Arm/Group | Pt 1: MK-3281 100 mg BID (Panel A) | Pt 1: MK-3281 200 mg BID (Panel B) | Pt 1: MK-3281 400 mg BID (Panel C) | Pt 1: MK-3281 800 mg BID (Panel D) | Pt 2: MK-3281 800 mg BID (Panel E) | Pt 2: MK-3281 800 mg BID (Panel F) | Pt 2: MK-3281 1200 mg BID (Panel G) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/3 | 0/14
Other Adverse Events (participants affected / at risk) | 5/7 | 3/6 | 4/6 | 5/6 | 3/6 | 12/12 | 2/3 | 12/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pt 1: MK-3281 100 mg BID (Panel A) (N=7) | Pt 1: MK-3281 200 mg BID (Panel B) (N=6) | Pt 1: MK-3281 400 mg BID (Panel C) (N=6) | Pt 1: MK-3281 800 mg BID (Panel D) (N=6) | Pt 2: MK-3281 800 mg BID (Panel E) (N=6) | Pt 2: MK-3281 800 mg BID (Panel F) (N=12) | Pt 2: MK-3281 1200 mg BID (Panel G) (N=3) | Placebo (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Catheter site haematoma (General disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device breakage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (5) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less